CLINICAL TRIAL: NCT05526183
Title: Phase I Randomized Double-Blind Clinical Trial With New SARS-CoV-2 CoVacHGMix Type 5 Adenoviral Vector Vaccine in Healthy Volunteers Aged 18-45 Years
Brief Title: Phase I Clinical Trial With New SARS-CoV-2 CoVacHGMix Type 5 Adenoviral Vector Vaccine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other); MonitorCRO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MON.760.159.3
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
Keywords: Vaccine-SARS-Cov-2-Adenoviral vector
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Parallel arm, double blind study with no control arm. Two doses of vaccine will be administered and the randomization will be performed for dose levels.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Vaccines will be provided to the study pharmacist and the randomization to dose levels will be prepared by the pharmacist. The vaccines will be provided to the investigators with volunteer numbers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose arm (Experimental): Low dose (5x1010 VP, i.m.); CoVacHGMix (with equal amounts of CoVacHGA1320, CoVacHGB420, CoVacHGC720 and CoVacHGD1480 adenoviral vector mix, as 0.5 solution) Intramuscular injection, two injections 28 days apart
  Interventions: Biological: Adeno-viral vector vaccine
- High dose arm (Experimental): High dose (1x1011 VP, i.m.); CoVacHGMix (with equal amounts of CoVacHGB420, CoVacHGC720 and CoVacHGD1480 adenoviral vector mix, as 1.0 solution) Intramuscular injections, two injections 28 days apart
  Interventions: Biological: Adeno-viral vector vaccine

INTERVENTIONS:
Biological: Adeno-viral vector vaccine — The vaccine will be injected intramuscularly, as two doses 28 days apart. Two different dosages will be given to volunteers (low dose: 5x1010 and high dose: 1x1011)

SUMMARY:
The CoVacHGMix adenoviral vector vaccine is a new vaccine developed to protect against SARS-CoV-2 and is a Phase I study designed based on adaptive clinical trial standards. In this Phase I study, it is aimed to test the safety and efficacy of the investigational product at 2 different dose levels (low: 5x1010 and high: 1x1011) in volunteers aged 18-59 years. Vaccination will be performed as two doses: on days 0 and 28. In line with adaptive design standards, Phase I will be transferred to Phase II. In this phase, 2 different dose levels will be tested, and the dose and application forms in Phase II will be determined according to the results of Phase I. One of the aims of the study is to collect sufficient data to determine the final dose and method of administration to be applied in the phase III study and clinic.

DETAILED DESCRIPTION:
The study is planned as a safety and immunogenicity efficacy study in healthy volunteers . Dose groups are as follows:

* Low Dose (2 injections 28 days apart): Treatment (n=18) CoVacHGMix (Adenoviral vector mix (0.5 mL) containing equal amounts of CoVacHGA1320, CoVacHGB420, CoVacHGC720 and CoVacHGD1480)
* High Dose (2 injections 28 days apart): Treatment (n=18) CoVacHGMix (adenoviral vector mix (1 mL) containing equal amounts of CoVacHGA1320, CoVacHGB420, CoVacHGC720, and CoVacHGD1480 After the first dose of vaccine (low dose group) was administered to the first two volunteers on day zero, no application will be made on the first day. On the second day, 1st dose of vaccine will be administered to 2 volunteers in the high dose group. Volunteers to be treated will remain in quarantine for 1 day before the application and will be monitored in the clinic for 24 hours after the application. Volunteers will be physically examined daily and blood samples will be taken for analysis. On the seventh day, the Independent Data Monitoring Committee (IDMC) will evaluate the clinical and laboratory data of the first 4 volunteers. Following the approval of the committee (Day 8), the first dose in all groups will continue to be freely available. On the 27th day, all volunteers who received their first dose of vaccines will be subjected to the PCR test and those who are negative according to the test results will be hospitalized for the administration of their second dose.

İe., On the 28th day, the first two volunteers from the low-dose group (two volunteers who received the low-dose vaccine on the first day) will be administered the 2nd dose of vaccine. On the thirtieth day, the first two volunteers from the high-dose group (two volunteers who received the high-dose vaccine on the first day) will be administered the 2nd vaccine dose. After the evaluation and approval of the clinical and laboratory data of the 4 volunteers whose second dose applications were completed by the safety committee, second dose administrations to the rest of volunteers will be continued from the 35th day.

ELIGIBILITY:
Inclusion Criteria:

I-1 Healthy volunteers of both sexes aged 18-59 years I-2 Able to give signed informed consent, I-3 Will be able to comply with the study protocol for approximately 6 months (depending on the group), I-4 HIV, Hepatitis B and C tests are negative, I-5 Body temperature below 37.2oC I-6 COVID-19 IgG and IgM antibodies negative and no history of symptomatic disease, I-7 Those who have not previously received any COVID-19 vaccines I-8 Negative qPCR SARS-CoV-2 result in nasopharynx or sputum samples, I-9 Body mass index between 18-35 kg/m2, I-10 Abnormal finding in complete blood count, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, urea, creatinine and fasting blood sugar between the normal reference values or detected in any laboratory parameter is Grade 1 according to the opinion of the investigator* volunteers not older (>Grade 1) I-11 Good general health (history and physical examination within 14 days prior to enrollment in the study), I-12 if female, healthy volunteers who are not pregnant or who can use appropriate contraception within 30 days before vaccine injection and within 6 months after vaccination will be included in the study.

I-13 Male volunteers who can use appropriate contraception within 6 months after vaccine injection will be included in the study.

Exclusion Criteria:

E-1. Subjects with a history of seizures, encephalopathy or psychosis, E-2. Subjects who have a known allergy to any vaccine or are allergic to any component of the vaccine to be administered, E-3. Pregnant or lactating women, women who have a positive pregnancy test or plan to become pregnant within the next 6 months.

E-4. Subjects whose body temperature is above 37.2oC at the time of vaccination or who have signs of active infection, E-5. Subjects with a positive history of SARS (SARS-CoV-1) (based on voluntary declaration), E-6.Subjects with severe cardiovascular disease (arrhythmia, conduction block, myocardial infarction, uncontrolled hypertension), E-7. Subjects with serious chronic diseases (asthma, diabetes, thyroid diseases, etc.), E-8. Subjects with congenital or acquired angioedema, E-9. Subjects with a diagnosis of immunodeficiency, E-10. Subjects with a diagnosis of bleeding diathesis, E-11. Subjects who take immunosuppressive treatment, those who take anti-allergic treatment, those who take cytotoxic treatment, those who take inhaled corticosteroids (except for allergic rhinitis or topical steroid ointments), E-12. Subjects who received blood and blood product transfusion in the last 4 months, E-13. Subjects who participated in any vaccine study or took experimental drugs within 1 month before starting the study, E-14. Subjects who received any live vaccines in the 1 month prior to the study E-15. Subjects who received inactivated vaccine within 14 days of starting the study E-16. Subjects receiving active tuberculosis treatment, E-17. Subjects with a personal or family history of thrombosis and thromboembolism, persons prone to thrombosis E-18. According to the researcher's evaluation, those who have any condition (medical, psychological, social, etc.) that may impair the volunteer's compliance with the study will be excluded from the study.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Day1 to 168 days after vaccination
  Adverse events

SECONDARY OUTCOMES:
Immunogenicity | 12 months
  Serum IgG and IgM titres (as compared to neutralizing antibody titres derived from convalescent plasma samples of patients).

CONTACTS AND LOCATIONS:
Overall Officials: Ekmel Olcay, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Bilkent, Ankara, Bilkent, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No